CLINICAL TRIAL: NCT00323622
Title: An Open Study for a 2-year Period to Confirm the Safety and Immunogenicity of the Candidate Malaria Vaccine RTS,S/AS02A in Mozambican Children Aged 1 to 4 Years at the Time of First Vaccine Dose.
Brief Title: Long-Term Follow-up of Children for a 2-Year Period to Confirm the Safety and Immunogenicity of GSK 257049 Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 104297
Record Dates: First submitted 2005-09-08; First posted 2006-05-09 (Estimated); Results first posted 2014-03-27 (Estimated); Last update posted 2016-12-09 (Estimated); Status verified 2016-10

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — RTS,S-AS02A vaccine; Hiberix; Heptavalent Pneumococcal Conjugate Vaccine; fanasil, pyrimethamine drug combination; Amodiaquine

ARMS (8):
- Cohort 1-RTS,S/AS02A <24M Group (Experimental): Subjects, male and female, aged 12 to 24 months at first vaccination, were administered 3 doses of RTS,S/AS02A (GSK 257049) vaccine at Months 0, 1 and 2 in the NCT00197041 Study. No additional dose of vaccine or drug was administered during this open follow-up NCT00323622 study. Subjects in this group are part of the Cohort 1 of the study, which was followed for analysis of malaria infection.
  Interventions: Biological: GSK Biologicals' candidate Plasmodium falciparum malaria vaccine 257049
- Cohort 1-RTS,S/AS02A ≥24M Group (Experimental): Subjects, male and female, aged between 24 and 48 months at first vaccination, were administered 3 doses of RTS,S/AS02A (GSK 257049) vaccine at Months 0, 1 and 2 in the NCT00197041 Study. No additional dose of vaccine or drug was administered during this open follow-up NCT00323622 study. Subjects in this group are part of the Cohort 1 of the study, which was followed for analysis of malaria infection.
  Interventions: Biological: GSK Biologicals' candidate Plasmodium falciparum malaria vaccine 257049
- Cohort 2-RTS,S/AS02A <24M Group (Experimental): Subjects, male and female, aged 12 to 24 months at first vaccination, were administered 3 doses of RTS,S/AS02A (GSK 257049) vaccine at Months 0, 1 and 2 in the NCT00197041 Study. Subjects in this group are part of the Cohort 2 of the study, which was followed for analysis of malaria disease. As Cohort 2 subjects, subjects in this group also received as part of the Primary NCT00197041 Study one dose of sulfadoxine-pyrimethamine and amodiaquine per day for 3 days 4 weeks prior to onset of surveillance, so as to clear any parasitemia. No additional dose of vaccine or drug was administered during this open follow-up NCT00323622 study.
  Interventions: Biological: GSK Biologicals' candidate Plasmodium falciparum malaria vaccine 257049; Drug: sulfadoxine-pyrimethamine; Drug: amodiaquine
- Cohort 2-RTS,S/AS02A ≥24M Group (Experimental): Subjects, male and female, aged between 24 and 48 months at first vaccination, were administered 3 doses of RTS,S/AS02A (GSK 257049) vaccine at Months 0, 1 and 2 of the NCT00197041 Study. Subjects in this group are part of the Cohort 2 of the study, which was followed for analysis of malaria disease. As Cohort 2 subjects, subjects in this group also received as part of the Primary NCT00197041 Study one dose of sulfadoxine-pyrimethamine and amodiaquine per day for 3 days 4 weeks prior to onset of surveillance, so as to clear any parasitemia. No additional dose of vaccine or drug was administered during this open follow-up NCT00323622 study.
  Interventions: Biological: GSK Biologicals' candidate Plasmodium falciparum malaria vaccine 257049; Drug: sulfadoxine-pyrimethamine; Drug: amodiaquine
- Cohort 1-Prevnar-Hiberix <24M Group (Active Comparator): Subjects, male and female, aged 12 to 24 months at first vaccination, were administered 2 doses of Prevnar™ vaccine at Months 0 and 2 and 1 dose of Hiberix® vaccine at Month 1 in the Primary NCT00197041 Study. No additional dose of vaccine or drug was administered during this open follow-up NCT00323622 study. Subjects in this group are part of the Cohort 1 of the study, which was followed for analysis of malaria infection.
  Interventions: Biological: Hiberix®; Biological: Prevnar™
- Cohort 1-Engerix-B ≥24M Group (Active Comparator): Subjects, male and female, aged between 24 and 48 months at first vaccination, were administered 3 doses of Engerix®-B vaccine at Months 0, 1 and 2 in the Primary NCT00197041 Study. No additional dose of vaccine or drug was administered during this open follow-up NCT00323622 study. Subjects in this group are part of the Cohort 1 of the study, which was followed for analysis of malaria infection.
  Interventions: Biological: Engerix™-B
- Cohort 2-Prevnar- Hiberix <24M Group (Active Comparator): Subjects, male and female, aged 12 to 24 months at first vaccination, were administered 2 doses of Prevnar™ vaccine at Months 0 and 2 and 1 dose of Hiberix® vaccine at Month 1 in the Primary NCT00197041 Study. Subjects in this group are part of the Cohort 2 of the study, which was followed for analysis of malaria disease. As Cohort 2 subjects, subjects in this group also received as part of the Primary NCT00197041 Study one dose of sulfadoxine-pyrimethamine and amodiaquine per day for 3 days 4 weeks prior to onset of surveillance, so as to clear any parasitemia. No additional dose of vaccine or drug was administered during this open follow-up NCT00323622 study.
  Interventions: Biological: Hiberix®; Biological: Prevnar™; Drug: sulfadoxine-pyrimethamine; Drug: amodiaquine
- Cohort 2-Engerix-B ≥24M Group (Active Comparator): Subjects, male and female, aged between 24 and 48 months at first vaccination, were administered 3 doses of Engerix®-B vaccine at Months 0, 1 and 2 in the Primary NCT00197041 Study. Subjects in this group are part of the Cohort 2 of the study, which was followed for analysis of malaria disease. As Cohort 2 subjects, subjects in this group also received as part of the Primary NCT00197041 Study one dose of sulfadoxine-pyrimethamine and amodiaquine per day for 3 days 4 weeks prior to onset of surveillance, so as to clear any parasitemia. No additional dose of vaccine or drug was administered during this open follow-up NCT00323622 study.
  Interventions: Biological: Engerix™-B; Drug: sulfadoxine-pyrimethamine; Drug: amodiaquine

INTERVENTIONS:
Biological: GSK Biologicals' candidate Plasmodium falciparum malaria vaccine 257049 — IM injection in the deltoid muscle
  Other Names: RTS; S/AS02A vaccine
  Arms: Cohort 1-RTS,S/AS02A <24M Group; Cohort 1-RTS,S/AS02A ≥24M Group; Cohort 2-RTS,S/AS02A <24M Group; Cohort 2-RTS,S/AS02A ≥24M Group
Biological: Engerix™-B — IM injection in the deltoid muscle
  Arms: Cohort 1-Engerix-B ≥24M Group; Cohort 2-Engerix-B ≥24M Group
Biological: Hiberix® — IM injection in the deltoid muscle
  Arms: Cohort 1-Prevnar-Hiberix <24M Group; Cohort 2-Prevnar- Hiberix <24M Group
Biological: Prevnar™ — IM injection in the deltoid muscle
  Arms: Cohort 1-Prevnar-Hiberix <24M Group; Cohort 2-Prevnar- Hiberix <24M Group
Drug: sulfadoxine-pyrimethamine — 1 dose orally per day for 3 days, 4 weeks prior to onset of surveillance
  Arms: Cohort 2-Engerix-B ≥24M Group; Cohort 2-Prevnar- Hiberix <24M Group; Cohort 2-RTS,S/AS02A <24M Group; Cohort 2-RTS,S/AS02A ≥24M Group
Drug: amodiaquine — 1 dose orally per day for 3 days, 4 weeks prior to onset of surveillance
  Arms: Cohort 2-Engerix-B ≥24M Group; Cohort 2-Prevnar- Hiberix <24M Group; Cohort 2-RTS,S/AS02A <24M Group; Cohort 2-RTS,S/AS02A ≥24M Group

SUMMARY:
The RTS,S/AS02A vaccine (or GSK 257049 vaccine), GSK Biologicals' candidate Plasmodium falciparum (P. falciparum) malaria vaccine is being developed for the routine immunization of infants and children living in malaria endemic areas. The vaccine would offer protection against malaria disease due to the parasite P. falciparum. The vaccine would also provide protection against infection with hepatitis B virus (HBV).

This phase IIb trial is being carried out following the demonstration of efficacy of the candidate malaria vaccine in children in Mozambique: there, the vaccine demonstrated approximately 30% efficacy against clinical episodes of malaria and approximately 58% efficacy against severe malaria disease.

In this study, the children from Mozambique (NCT= NCT00197041) are followed-up to assess the safety, immunogenicity and efficacy of the candidate malaria vaccine for a two year period commencing 21 months after Dose 1.

This protocol posting deals with objectives & outcome measures of the extension phase at year 2. During this extension study, no new subjects will be recruited and no vaccine will be administered.

The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

ELIGIBILITY:
Inclusion criteria:

* Completion of Visit 7, Month 21 of 104297 (NCT= NCT00197041).
* Written informed consent obtained from the parent(s) or guardian(s) of the subject

Exclusion criteria:

* Planned use of any investigational or non-registered drug or vaccine during the study period.
* Simultaneous participation in any other clinical trial

Ages: 33 Months to 69 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1737 (Actual)
Dates: Start 2005-04; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Maputo, Mozambique

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Alonso PL, Sacarlal J, Aponte JJ, Leach A, Macete E, Aide P, Sigauque B, Milman J, Mandomando I, Bassat Q, Guinovart C, Espasa M, Corachan S, Lievens M, Navia MM, Dubois MC, Menendez C, Dubovsky F, Cohen J, Thompson R, Ballou WR. Duration of protection with RTS,S/AS02A malaria vaccine in prevention of Plasmodium falciparum disease in Mozambican children: single-blind extended follow-up of a randomised controlled trial. Lancet. 2005 Dec 10;366(9502):2012-8. doi: 10.1016/S0140-6736(05)67669-6. PMID 16338450
- [Background] Aponte et al. A 4 years follow-up of the safety, immunogenicity and efficacy of the candidate malaria vaccine RTS,S/AS02A in children vaccinated at aged 1 to 4 years in a malaria-endemic region of Mozambique. Abstract presented at the 56th Annual Meeting ASTMH, Philadelphia, PA, USA, 05-07 November 2007.
- [Background] Sacarlal J, Aide P, Aponte JJ, Renom M, Leach A, Mandomando I, Lievens M, Bassat Q, Lafuente S, Macete E, Vekemans J, Guinovart C, Sigauque B, Sillman M, Milman J, Dubois MC, Demoitie MA, Thonnard J, Menendez C, Ballou WR, Cohen J, Alonso PL. Long-term safety and efficacy of the RTS,S/AS02A malaria vaccine in Mozambican children. J Infect Dis. 2009 Aug 1;200(3):329-36. doi: 10.1086/600119. PMID 19569964
- [Derived] Aide P, Dobano C, Sacarlal J, Aponte JJ, Mandomando I, Guinovart C, Bassat Q, Renom M, Puyol L, Macete E, Herreros E, Leach A, Dubois MC, Demoitie MA, Lievens M, Vekemans J, Loucq C, Ballou WR, Cohen J, Alonso PL. Four year immunogenicity of the RTS,S/AS02(A) malaria vaccine in Mozambican children during a phase IIb trial. Vaccine. 2011 Aug 11;29(35):6059-67. doi: 10.1016/j.vaccine.2011.03.041. Epub 2011 Apr 7. PMID 21443960
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 104297 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 104297 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 104297 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 104297 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 104297 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 104297 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This current study NCT00323622, a follow-up (FU) study to the primary study NCT00197041, is aimed at vaccine safety assessment, and took place from Months 21 to 45 (Month 0 = Dose 1 administration of RTS,S/AS02A (GSK 257049) or comparator vaccine in the primary study).
Pre-assignment Details: Once re-enrolled, subjects in this study were allocated to the same groups as in the NCT00197041 study, as well as the same cohorts, e. a. Cohorts 1 and 2 whose subjects were followed for analysis of, respectively, malaria infection and disease.
Groups:
- Cohort 1-RTS,S/AS02A<24M Group: Subjects, male and female, aged 12 to 24 months at first vaccination, were administered 3 doses of RTS,S/AS02A (GSK 257049) vaccine at Months 0, 1 and 2 in the NCT00197041 Study. No additional dose of vaccine or drug was administered during this open follow-up NCT00323622 study. Subjects in this group are part of the Cohort 1 of the study, which was followed for analysis of malaria infection
- Cohort 1-RTS,S/AS02A≥24M Group: Subjects, male and female, aged between 24 and 48 months at first vaccination, were administered 3 doses of RTS,S/AS02A (GSK 257049) vaccine at Months 0, 1 and 2 in the NCT00197041 Study. No additional dose of vaccine or drug was administered during this open follow-up NCT00323622 study. Subjects in this group are part of the Cohort 1 of the study, which was followed for analysis of malaria infection.
- Cohort 2-RTS,S/AS02A<24M Group: Subjects, male and female, aged 12 to 24 months at first vaccination, were administered 3 doses of RTS,S/AS02A (GSK 257049) vaccine at Months 0, 1 and 2 in the NCT00197041 Study. Subjects in this group are part of the Cohort 2 of the study, which was followed for analysis of malaria disease. As Cohort 2 subjects, subjects in this group also received as part of the Primary NCT00197041 Study one dose of sulfadoxine-pyrimethamine and amodiaquine per day for 3 days 4 weeks prior to onset of surveillance, so as to clear any parasitemia. No additional dose of vaccine or drug was administered during this open follow-up NCT00323622 study.
- Cohort 2-RTS,S/AS02A≥24M Group: Subjects, male and female, aged between 24 and 48 months at first vaccination, were administered 3 doses of RTS,S/AS02A (GSK 257049) vaccine at Months 0, 1 and 2 of the NCT00197041 Study. Subjects in this group are part of the Cohort 2 of the study, which was followed for analysis of malaria disease. As Cohort 2 subjects, subjects in this group also received as part of the Primary NCT00197041 Study one dose of sulfadoxine-pyrimethamine and amodiaquine per day for 3 days 4 weeks prior to onset of surveillance, so as to clear any parasitemia. No additional dose of vaccine or drug was administered during this open follow-up NCT00323622 study.
Period: Overall Study
Arm/Group | Cohort 1-RTS,S/AS02A<24M Group | Cohort 1-RTS,S/AS02A≥24M Group | Cohort 2-RTS,S/AS02A<24M Group | Cohort 2-RTS,S/AS02A≥24M Group | Cohort 1-Prevnar-Hiberix <24M Group | Cohort 1-Engerix-B ≥24M Group | Cohort 2-Prevnar- Hiberix <24M Group | Cohort 2-Engerix-B ≥24M Group
Started | 176 | 515 | 42 | 134 | 159 | 528 | 43 | 140
Completed | 145 | 423 | 38 | 122 | 120 | 454 | 38 | 125
Not Completed | 31 | 92 | 4 | 12 | 39 | 74 | 5 | 15
Not completed — Other | 30 | 91 | 4 | 12 | 32 | 74 | 5 | 13
Not completed — Death | 1 | 1 | 0 | 0 | 7 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1-RTS,S/AS02A <24M Group | Cohort 1-RTS,S/AS02A ≥24M Group | Cohort 2-RTS,S/AS02A <24M Group | Cohort 2-RTS,S/AS02A ≥24M Group | Cohort 1-Prevnar-Hiberix <24M Group | Cohort 1-Engerix-B ≥24M Group | Cohort 2-Prevnar- Hiberix <24M Group | Cohort 2-Engerix-B ≥24M Group | Total
Number analyzed (Participants) | 176 | 515 | 42 | 134 | 159 | 528 | 43 | 140 | 1737
Age, Continuous [Mean (Standard Deviation); unit: Months] | 38 (4.0) | 62 (11.0) | 39 (4.0) | 62 (9.0) | 38 (3.0) | 62 (10.0) | 38 (3.0) | 61 (9.0) | 50.0 (6.6)
Gender [Count of Participants; unit: Participants]
  Female | 85 | 240 | 19 | 67 | 79 | 252 | 16 | 78 | 836
  Male | 91 | 275 | 23 | 67 | 80 | 276 | 27 | 62 | 901

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: Throughout the entire study period: from Month 21 to Month 45 (Month 0 = administration of Dose 1 of RTS,S/AS02A or comparator vaccine in the NCT00197041 study).
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects vaccinated in the primary NCT00197041 study, and re- enrolled in this follow-up NCT 00323622 study, and for whom data were available.
Measure: Number; unit: Subjects
Arm/Group | Cohort 1-RTS,S/AS02A <24M Group | Cohort 1-RTS,S/AS02A ≥24M Group | Cohort 2-RTS,S/AS02A <24M Group | Cohort 2-RTS,S/AS02A ≥24M Group | Cohort 1-Prevnar-Hiberix <24M Group | Cohort 1-Engerix-B ≥24M Group | Cohort 2-Prevnar- Hiberix <24M Group | Cohort 2-Engerix-B ≥24M Group
Number analyzed (Participants) | 176 | 515 | 42 | 134 | 159 | 528 | 43 | 140
Subjects | 21 | 17 | 1 | 0 | 24 | 29 | 1 | 4

2. Secondary Outcome: Anti-circumsporozoite Protein (CS) Antibody Concentrations.
Description: Concentrations for anti-CS antibodies are presented as Geometric Mean Concentrations (GMCs), expressed in Enzyme-Linked Immunosorbent Assay (ELISA) units per milliliter (EL.U/mL). The cut-off of the assay was the seropositivity cut-off of 0.5 EL.U/mL. Subjects were pooled across age ranges for this outcome measure.
Time Frame: At Months 33 and 45 (Month 0 = administration of Dose 1 of RTS,S/AS02A or comparator vaccine in the NCT00197041 study).
Population: The Long Term According-to-Protocol (ATP) cohort for immunogenicity included all enrolled subjects from the primary study ATP cohort for immunogenicity who did not receive any additional vaccine dose containing circumsporozoite protein or hepatitis B antigens, with blood sample within protocol-defined time limits and available antibody measurements
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Groups:
- Cohort 1-RTS,S/AS02A Group: Subjects, male and female, aged between 12 and 48 months at the time of the first vaccination, were administered 3 doses of RTS,S/AS02A (GSK 257049) vaccine at Months 0, 1 and 2 in the NCT00197041 Study. No additional dose of vaccine or drug was administered during this open follow-up NCT00323622 study. This group is part of the Cohort 1 of the study, which was followed for analysis of malaria infection, and pools subjects from the Cohort 1-RTS,S/AS02A Cohort 1-RTS,S/AS02A <24M and Cohort 1-RTS,S/AS02A ≥24M groups.
- Cohort 1-Engerix-B/Prevnar-Hiberix Group: Subjects, male and female, aged 12 up to 24 months at first vaccination, were administered 2 doses of Prevnar™ vaccine at Months 0 and 2 and 1 dose of Hiberix® vaccine at Month 1 in the Primary NCT00197041 Study. Subjects, male and female, aged between 24 and 48 months first vaccination, were administered 3 doses of Engerix®-B vaccine at Months 0, 1 and 2 in the Primary NCT00197041 Study. No additional dose of vaccine or drug was administered during this open follow-up NCT00323622 study. This group is part of the Cohort 1 of the study, which was followed for analysis of malaria infection, and pools subjects from the Cohort 1-Engerix-B ≥24M and Cohort 1-Prevnar-Hiberix <24M groups.
- Cohort 2-RTS,S/AS02A Group: Subjects, male and female, aged between 12 and 48 months at the time of the first vaccination, were administered 3 doses of RTS,S/AS02A (GSK 257049) vaccine at Months 0, 1 and 2 in the NCT00197041 Study. This group is part of the Cohort 2 of the study, which was followed for analysis of malaria disease, and pools subjects from the Cohort 2-RTS,S/AS02A <24M and Cohort 2-RTS,S/AS02A ≥24M groups. As Cohort 2 subjects, subjects in this group also received as part of the Primary NCT00197041 Study one dose of sulfadoxine-pyrimethamine and amodiaquine per day for 3 days 4 weeks prior to onset of surveillance, so as to clear any parasitemia. No additional dose of vaccine or drug was administered during this open follow-up NCT00323622 study.
- Cohort 2-Engerix-B/Prevnar-Hiberix Group: Subjects, male and female, aged 12 to 24 months at first vaccination, were administered 2 doses of Prevnar™ vaccine at Months 0 and 2 and 1 dose of Hiberix® vaccine at Month 1 in the Primary NCT00197041 Study. Subjects, male and female, aged between 24 and 48 months at first vaccination, were administered 3 doses of Engerix®-B vaccine at Months 0, 1 and 2 in the Primary NCT00197041 Study. This group is part of the Cohort 2 of the study, which was followed for analysis of malaria disease, and pools subjects from the Cohort 2-Engerix-B ≥24M and Cohort 2-Prevnar-Hiberix <24M groups. As Cohort 2 subjects, subjects in this group also received as part of the Primary NCT00197041 Study one dose of sulfadoxine-pyrimethamine and amodiaquine per day for 3 days 4 weeks prior to onset of surveillance, so as to clear any parasitemia. No additional dose of vaccine or drug was administered during this open follow-up NCT00323622 study.
Arm/Group | Cohort 1-RTS,S/AS02A Group | Cohort 1-Engerix-B/Prevnar-Hiberix Group | Cohort 2-RTS,S/AS02A Group | Cohort 2-Engerix-B/Prevnar-Hiberix Group
Number analyzed (Participants) | 490 | 487 | 150 | 149
EL.U/mL
  Month 33 [N = 490, 487, 149, 149] | 10.1 [8.9 to 11.4] | NA [NA to NA] — GMC were not calculated as concentration fell below the assay cut-off | 16.2 [13.1 to 20.0] | 0.6 [0.5 to 0.7]
  Month 45 [N = 452, 447, 150, 145] | 8.9 [7.8 to 10.1] | NA [NA to NA] — GMC were not calculated as concentration fell below the assay cut-off | 15.4 [12.7 to 18.6] | 0.4 [0.4 to 0.5]

3. Secondary Outcome: Anti-hepatitis B (HBs) Antibody Concentrations.
Description: Concentrations are presented as geometric mean concentrations (GMCs), expressed in milli-international units per milliliter (mIU/mL). Anti-HBs antibody concentration levels were measured in blood samples from Cohort 2 only.
Time Frame: At Months 33 and 45 (Month 0 = administration of Dose 1 of RTS,S/AS02A or comparator vaccine in the NCT00197041 study).
Population: The Long Term According-to-Protocol (ATP) cohort for immunogenicity included all enrolled subjects from the primary study ATP cohort for immunogenicity who did not receive any additional vaccine dose containing circumsporozoite protein or hepatitis B antigens,with blood sample within protocol-defined time limits and available antibody measurements.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Cohort 2-RTS,S/AS02A <24M Group | Cohort 2-RTS,S/AS02A ≥24M Group | Cohort 2-Prevnar- Hiberix <24M Group | Cohort 2-Engerix-B ≥24M Group
Number analyzed (Participants) | 35 | 116 | 34 | 115
mIU/mL
  Month 33 [N = 33, 116, 34, 115] | 4008.6 [2266.7 to 7089.1] | 1842.5 [1413.7 to 2401.3] | 20.3 [10.9 to 37.9] | 67.4 [47.5 to 95.7]
  Month 45 [N = 35, 115, 32, 113] | 3323.8 [1908.4 to 5788.8] | 1557.0 [1187.6 to 2041.4] | 26.6 [13.0 to 54.1] | 99.4 [73.1 to 135.1]

4. Secondary Outcome: Time to First or Only Clinical Episode of Symptomatic Plasmodium Falciparum Malaria Infection (PFMI) of Primary Case Definition
Description: Malaria infection by Plasmodium falciparum was detected by passive case detection. A symptomatic PFMI episode of Primary Case Definition (PCD) was defined as the presence of P. falciparum asexual parasitaemia above 2500 per µL on Giemsa stained thick blood films accompanied by fever (axillary temperature equal or above 37.5 degrees Celsius at the time of presentation) occurring in an unwell child brought for treatment to a healthcare facility. The time to first or only episode of symptomatic PFMI is expressed in terms of rate of first PFMI (RPFMI), that is, the number of PFMI events reported (n) over the period elapsed until the PFMI event occurred (i.e. events per Persons Year at Risk [PYAR]) for each group. Analysis for this outcome was solely performed on Cohort 1 subjects, with groups pooled across age ranges.
Time Frame: From Month 21 to Month 33 (M21-33), and from Month 33 to Month 45 (M33-45). Month 0 = administration of Dose 1 of RTS,S/AS02A or comparator vaccine in study NCT00197041
Population: The analysis was performed on the According-to-Protocol cohort for efficacy, which included all evaluable subjects who had received the 3 doses of the RTS,S/AS02 or control vaccine(s) in the Primary NCT00197041, and with available data concerning efficacy measures starting 14 days post Dose 3 of RTS,S/AS02A or comparator vaccine(s).
Measure: Number; unit: n/PYAR
Arm/Group | Cohort 1-RTS,S/AS02A Group | Cohort 1-Engerix-B/Prevnar-Hiberix Group
Number analyzed (Participants) | 650 | 645
n/PYAR
  RPFMI - PCD - M21-33 (N=650;645) | 0.330 | 0.375
  RPFMI - PCD - M33-45 (N=638;629) | 0.140 | 0.149
Statistical Analysis 1: Comparison: Cohort 1-RTS,S/AS02A Group vs Cohort 1-Engerix-B/Prevnar-Hiberix Group; The analysis aimed to compare rates of first PFMI (RPFMI) between groups over the Months 21-33 time period. Using RFPMI, a Cox model was used to evaluate vaccine efficacy (VE) allowing for adjustment factors. VE, point estimate of efficacy adjusted for covariates, was calculated as 1 - (minus) [Hazard Ratio (HR) in Cohort 1 - GSK RTS,S/AS02A Group [HR1]) divided by HR in Cohort 1 - Engerix-B/Prevnar-Hiberix Group [HR2])], i. e. 1 - (HR1/HR2); Test type: Superiority or Other; p = 0.08, Regression, Cox — The p-value presented is the Wald Chi-square p-value from the Cox regression model; Point estimate of efficacy was adjusted for age, geographical area of residence, bednet use and distance from health center; 1 - (HR1/HR2) = 16.8, 95% CI 2-sided [-2.50 to 32.40]
Statistical Analysis 2: Comparison: Cohort 1-RTS,S/AS02A Group vs Cohort 1-Engerix-B/Prevnar-Hiberix Group; The analysis aimed to compare rates of first PFMI (RPFMI) between groups over the Months 33-45 time period. Using RFPMI, a Cox model was used to evaluate vaccine efficacy (VE) allowing for adjustment factors. VE, point estimate of efficacy adjusted for covariates, was calculated as 1 - (minus) [Hazard Ratio (HR) in Cohort 1 - RTS,S/AS02A Group [HR1]) divided by HR in Cohort 1 - Engerix-B/Prevnar-Hiberix Group [HR2])], i. e. 1 - (HR1/HR2); Test type: Superiority or Other; p = 0.43, Regression, Cox — The p-value presented is the Wald Chi-square p-value from the Cox regression model; [statistical method as in outcome 4, analysis 1]; 1 - (HR1/HR2) = 11.8, 95% CI 2-sided [-20.11 to 35.18]

5. Secondary Outcome: Time to First or Only Episode of Symptomatic Plasmodium Falciparum Malaria Infection (PFMI) of Secondary Case Definition 1
Description: PFMI was detected by passive case detection. Symptomatic PFMI of Secondary Case Definition (SCD) 1 was defined as the presence of P. falciparum asexual parasitaemia (any level if parasitemia) on Giemsa stained thick blood films accompanied by fever (axillary temperature equal or above 37.5 degrees Celsius) in an unwell child brought for treatment. The time to first or only episode of symptomatic PFMI is expressed in terms of rate of first PFMI (RPFMI), that is, the number of PFMI events reported (n) over the period elapsed until the PFMI event occurred (i.e. events per Persons Year at Risk [PYAR]) for each group. Analysis for this outcome was solely performed on Cohort 1 subjects, with groups pooled across age ranges.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Number; unit: n/PYAR
Arm/Group | Cohort 1-RTS,S/AS02A Group | Cohort 1-Engerix-B/Prevnar-Hiberix Group
Number analyzed (Participants) | 650 | 645
n/PYAR
  RPFMI - SCD 1 - M21-33 (N=650;645) | 0.365 | 0.409
  RPFMI - SCD 1 - M33-45 (N=638;629) | 0.161 | 0.174
Statistical Analysis 1: Comparison: Cohort 1-RTS,S/AS02A Group vs Cohort 1-Engerix-B/Prevnar-Hiberix Group; The analysis aimed to compare rates of first PFMI (RPFMI) between groups over the Months 21-33 time period. Using RFPMI, a Cox model was used to evaluate vaccine efficacy (VE) allowing for adjustment factors. VE, point estimate of efficacy adjusted for covariates, was calculated as 1 - (minus) [Hazard Ratio (HR) in Cohort 1 - RTS,S/AS02A Group [HR1]) divided by HR in Cohort 1 - Engerix-B/Prevnar-Hiberix Group [HR2])], i. e. 1 - (HR1/HR2); Test type: Superiority or Other; p = 0.11, Regression, Cox — The p-value presented is the Wald Chi-square p-value from the Cox regression model; [statistical method as in outcome 4, analysis 1]; 1 - (R1/R2) = 14.90, 95% CI 2-sided [-3.88 to 30.28]
Statistical Analysis 2: Comparison: Cohort 1-RTS,S/AS02A Group vs Cohort 1-Engerix-B/Prevnar-Hiberix Group; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p = 0.35, Regression, Cox — The p-value presented is the Wald Chi-square p-value from the Cox regression model; [statistical method as in outcome 4, analysis 1]; 1 - (R1/R2) = 12.79, 95% CI 2-sided [-16.27 to 34.59]

6. Secondary Outcome: Time to First or Only Episode of Symptomatic Plasmodium Falciparum Malaria Infection (PFMI) of Secondary Case Definition 2
Description: PFMI was detected by passive case detection. Symptomatic PFMI of Secondary Case Definition (SCD) 2 was defined as the presence of P. falciparum asexual parasitaemia (any level if parasitemia) on Giemsa stained thick blood films in an unwell child brought for treatment with a history of fever (axillary temperature equal or above 37.5 degrees Celsius) within 24 hours or documented fever. The time to first or only episode of symptomatic PFMI is expressed in terms of rate of first PFMI (RPFMI), that is, the number of PFMI events reported (n) over the period elapsed until the PFMI event occurred (i.e. events per Persons Year at Risk [PYAR]) for each group. Analysis for this outcome was performed on Cohort 1 subjects, with groups pooled across age ranges.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Number; unit: n/PYAR
Arm/Group | Cohort 1-RTS,S/AS02A Group | Cohort 1-Engerix-B/Prevnar-Hiberix Group
Number analyzed (Participants) | 650 | 645
n/PYAR
  RPFMI - SCD 2 - M21-33 (N=650;645) | 0.540 | 0.630
  RPFMI - SCD 2 - M33-45 (N=638;629) | 0.260 | 0.270
Statistical Analysis 1: Comparison: Cohort 1-RTS,S/AS02A Group vs Cohort 1-Engerix-B/Prevnar-Hiberix Group; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.01, Regression, Cox — The p-value presented is the Wald Chi-square p-value from the Cox regression model; [statistical method as in outcome 4, analysis 1]; 1 - (R1/R2) = 19.42, 95% CI 2-sided [4.62 to 31.93]
Statistical Analysis 2: Comparison: Cohort 1-RTS,S/AS02A Group vs Cohort 1-Engerix-B/Prevnar-Hiberix Group; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p = 0.54, Regression, Cox — The p-value presented is the Wald Chi-square p-value from the Cox regression model; 1 - (R1/R2) = 7.08, 95% CI 2-sided [-17.37 to 26.44]

7. Secondary Outcome: Time to First or Only Episode of Symptomatic Plasmodium Falciparum Malaria Infection (PFMI) of Secondary Case Definition 3
Description: PFMI was detected by passive case detection. Symptomatic PFMI of Secondary Case Definition (SCD) 3 was defined as the presence of P. falciparum asexual parasitaemia above 15000 per microliter (µL) on Giemsa stained thick blood films accompanied by fever (axillary temperature equal or above 37.5 degrees Celsius) in an unwell child brought for treatment to a healthcare facility. The time to first or only episode of symptomatic PFMI is expressed in terms of rate of first PFMI (RPFMI), that is, the number of PFMI events reported (n) over the period elapsed until the PFMI event occurred (i.e. events per Persons Year at Risk [PYAR]) for each group. Analysis for this outcome was performed on Cohort 1 subjects solely, with groups pooled across age ranges.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Number; unit: n/PYAR
Arm/Group | Cohort 1-RTS,S/AS02A Group | Cohort 1-Engerix-B/Prevnar-Hiberix Group
Number analyzed (Participants) | 650 | 645
n/PYAR
  RPFMI - SCD 3 - M21-33 (N=650;645) | 0.288 | 0.329
  RPFMI - SCD 3 - M33-45 (N=638;629) | 0.122 | 0.122
Statistical Analysis 1: Comparison: Cohort 1-RTS,S/AS02A Group vs Cohort 1-Engerix-B/Prevnar-Hiberix Group; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.10, Regression, Cox — The p-value presented is the Wald Chi-square p-value from the Cox regression model; 1 - (R1/R2) = 16.79, 95% CI 2-sided [-3.75 to 33.25]
Statistical Analysis 2: Comparison: Cohort 1-RTS,S/AS02A Group vs Cohort 1-Engerix-B/Prevnar-Hiberix Group; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p = 0.70, Regression, Cox — The p-value presented is the Wald Chi-square p-value from the Cox regression model; [statistical method as in outcome 4, analysis 1]; 1 - (R1/R2) = 6.31, 95% CI 2-sided [-31.00 to 32.99]

8. Secondary Outcome: Number of Primary Case Definition Clinical Episodes of Symptomatic Plasmodium Falciparum Malaria Infection (PFMI)
Description: PFMI was detected by passive case detection. A symptomatic PFMI episode of Primary Case Definition (PCD) was defined as the presence of P. falciparum asexual parasitaemia above 2500 per µL on Giemsa stained thick blood films accompanied by fever (axillary temperature equal or above 37.5 degrees Celsius at the time of presentation) occurring in an unwell child brought for treatment to a healthcare facility. The number of PFMI episodes (EPFMI) per person-year (pyr) was tabulated, using as unit EPFMI episode per pyr. Analysis for this outcome was performed on Cohort 1 subjects solely, with groups pooled across age ranges.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Number; unit: EPFMI episode per pyr
Arm/Group | Cohort 1-RTS,S/AS02A Group | Cohort 1-Engerix-B/Prevnar-Hiberix Group
Number analyzed (Participants) | 650 | 645
EPFMI episode per pyr
  EPFMI - PCD - M21-33 (N=650;645) | 252 | 291
  EPFMI - PCD - M33-45 (N=638;629) | 99 | 100

9. Secondary Outcome: Number of Subjects With Anemia.
Description: Anemia was indicated by a hematocrit level (HL) below (<) 25%. The numbers of subjects with HL below (<) and above or equal (≥) 25 %, and with missing HL results were tabulated. In the tabulation below, the number of subjects falling into the "HL ≥25%" category corresponds to the number of subjects with anemia as asked per outcome. Analysis for this outcome was performed on Cohort 1 subjects solely, with groups pooled across age ranges.
Time Frame: At Months 33 and 45 (Month 0 = administration of Dose 1 of RTS,S/AS02A or comparator vaccine in the NCT00197041 study).
Population: as for outcome 4
Measure: Number; unit: Subjects
Arm/Group | Cohort 1-RTS,S/AS02A Group | Cohort 1-Engerix-B/Prevnar-Hiberix Group
Number analyzed (Participants) | 650 | 645
Subjects
  HL <25%, Month 33 (N = 650, 645) | 2 | 2
  HL ≥25%, Month 33 (N = 650, 645]) | 584 | 593
  Missing Results, Month 33 (N = 650;645) | 64 | 50
  HL <25%, Month 45 (N = 638, 629) | 0 | 0
  HL ≥25%, Month 45 (N = 638, 629) | 540 | 543
  Missing Results, Month 45 (N = 638;629) | 98 | 86

10. Secondary Outcome: Number of Subjects Prevalent for Plasmodium Falciparum (P. Falciparum) Parasitemia
Description: Subjects prevalent for P. falciparum parasitemia were defined as subjects with the presence of P. falciparum asexual parasitemia above 0 per microliter (µL) on Giemsa stained thick blood films.Analysis for this outcome was performed on Cohort 1 subjects solely, with groups pooled across age ranges.
Time Frame: At Months 33 (M33) and 45 (M45) (Month 0 = administration of Dose 1 of RTS,S/AS02A or comparator vaccine in the NCT00197041 study).
Population: as for outcome 4
Measure: Number; unit: Subjects
Arm/Group | Cohort 1-RTS,S/AS02A Group | Cohort 1-Engerix-B/Prevnar-Hiberix Group
Number analyzed (Participants) | 590 | 596
Subjects
  Subjects prevalent for parasitemia, M33[N=590,590] | 93 | 121
  Subjects prevalent for parasitemia, M45[N=541,547] | 66 | 101

ADVERSE EVENTS:
Time Frame: SAE reports were collected from 21 to 45 months post Dose 1 of either vaccine.
Description: No reports of solicited symptoms or unsolicited AEs were collected during this study. Fatal SAEs were reported for a total of 11 subjects (1 in the Cohort 1-RTS,S/AS02A <24M Group, 1 in the Cohort 1-RTS,S/AS02A ≥24M Group, 7 in the Cohort 1-Prevnar-Hiberix <24M Group and 2 in the Cohort 2-Engerix-B ≥24M Group)
Arm/Group | Cohort 1-RTS,S/AS02A <24M Group | Cohort 1-RTS,S/AS02A ≥24M Group | Cohort 2-RTS,S/AS02A <24M Group | Cohort 2-RTS,S/AS02A ≥24M Group | Cohort 1-Prevnar-Hiberix <24M Group | Cohort 1-Engerix-B ≥24M Group | Cohort 2-Prevnar- Hiberix <24M Group | Cohort 2-Engerix-B ≥24M Group
Serious Adverse Events (participants affected / at risk) | 21/176 | 17/515 | 1/42 | 0/134 | 24/159 | 29/528 | 1/43 | 4/140
Other Adverse Events (participants affected / at risk) | 0/176 | 0/515 | 0/42 | 0/134 | 0/159 | 0/528 | 0/43 | 0/140
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1-RTS,S/AS02A <24M Group (N=176) | Cohort 1-RTS,S/AS02A ≥24M Group (N=515) | Cohort 2-RTS,S/AS02A <24M Group (N=42) | Cohort 2-RTS,S/AS02A ≥24M Group (N=134) | Cohort 1-Prevnar-Hiberix <24M Group (N=159) | Cohort 1-Engerix-B ≥24M Group (N=528) | Cohort 2-Prevnar- Hiberix <24M Group (N=43) | Cohort 2-Engerix-B ≥24M Group (N=140)
Ascariasis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Brain contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 — This SAE was fatal for one subject in the Cohort 1-Prevnar-Hiberix <24M Group.
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Encephalitis viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemophilus sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaria (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 — This SAE was fatal for one subject in the Cohort 1-Prevnar-Hiberix <24M Group.
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Pneumococcal sepsis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tinea capitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — This SAE was fatal for one subject in the Cohort 1-Prevnar-Hiberix <24M Group.
Cellulitis orbital (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cerebral malaria (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — This SAE was fatal for one subject in the Cohort 1-Prevnar-Hiberix <24M Group.
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Death (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Febrile convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 5 | 7 | 1 | 1
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 — This SAE was fatal for one subject in the Cohort 1-Prevnar-Hiberix <24M Group.
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Immunosuppression (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — This SAE was fatal for one subject in the Cohort 1-Prevnar-Hiberix <24M Group.
Kwashiorkor (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — This SAE was fatal for one subject in the Cohort 1-Prevnar-Hiberix <24M Group.
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — This SAE was fatal for one subject in the Cohort 1-Prevnar-Hiberix <24M Group.
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — This SAE was fatal for one subject in the Cohort 1-Prevnar-Hiberix <24M Group.
Pyoderma (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Salmonella sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 — This SAE was fatal for one subject in the Cohort 1-Prevnar-Hiberix <24M Group.
Streptococcal bacteremia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 — This SAE was fatal for one subject in the Cohort 1-Prevnar-Hiberix <24M Group and one subject in the Cohort 2-Engerix-B ≥24M Group
Underweight (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acquired immunodeficiency syndrome (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 — This SAE was fatal for 2 subjects in the Cohort 1-Prevnar-Hiberix <24M Group.
Anemia (Blood and lymphatic system disorders) | 12 | 8 | 1 | 0 | 14 | 9 | 0 | 1 — This SAE was fatal for one subject in the Cohort 1-RTS,S/AS02A <24M Group, one subject in the Cohort 1-RTS,S/AS02A ≥24M Group, and 3 subjects in the Cohort 1-Prevnar-Hiberix <24M Group
HIV Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — This SAE was fatal for one subject in the Cohort 1-RTS,S/AS02A ≥24M Group.
Plasmodium falciparum infection (Infections and infestations) | 20 | 14 | 1 | 0 | 18 | 19 | 1 | 2 — Occurrences of this SAE were fatal for one subject in the Cohort 1-RTS,S/AS02A <24M Group, one subject in the Cohort 1-RTS,S/AS02A ≥24M Group and 2 subjects in the Cohort 1-Prevnar-Hiberix <24M Group
Pneumonia (Infections and infestations) | 2 | 2 | 0 | 0 | 3 | 3 | 0 | 0 — This SAE was fatal for one subject in the Cohort 1-RTS,S/AS02A ≥24M Group and 3 subjects in the Cohort 1-Prevnar-Hiberix <24M Group.
Marasmus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — This SAE was fatal for one subject in the Cohort 1-RTS,S/AS02A ≥24M Group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.